CLINICAL TRIAL: NCT05878535
Title: The Efficacy And Safety Of Metformin For The Treatment Of Atrial Fibrillation
Brief Title: METFORMIN FOR ATRIAL FIBRILLATION
Acronym: MAFT
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Arab Contractors Medical Centre (Other)
Responsible Party: Principal Investigator, Eslam Abbas, MBChB, MSc, Principal Invstigator, Arab Contractors Medical Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: #18101829
Record Dates: First submitted 2023-05-18; First posted 2023-05-26 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2024-01

CONDITIONS: Atrial Fibrillation
Keywords: Atrial Fibrillation, metformin, MACE.
MeSH Terms: conditions — Atrial Fibrillation | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- The Metformin Group (MG) (Active Comparator): The group (n=385) will receive metformin oral tablets in addition to the standard rate/rhythm control strategy and anticoagulation.
  • Drug: metformin 850 mg oral tablets. Prescribed: Once daily PO with meals and 200 mL of water. The dose can be up-titrated to 1500-2000 mg divided q8-12hr with meals in enrolled diabetic patients as a monotherapy or combined with sulfonylurea.
  Other Name: Glucophage.
  Interventions: Drug: Metformin
- The Placebo Control Group (PCG) (Placebo Comparator): The group (n=385) will receive placebo oral tablets in addition to the standard rate/rhythm control strategy and anticoagulation.
  • Drug: Placebo oral tablets. Prescribed: Once daily PO with meals and 200 mL of water. Other Name: Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Metformin — Metformin 850 mg oral tablets. Prescribed: Once daily PO with meals and 200 mL of water. The dose can be up-titrated to 1500-2000 mg divided q8-12hr with meals in enrolled diabetic patients as a monotherapy or combined with sulfonylurea.
  Other Names: Glucophage, Glumetza, and Riomet.
  Arms: The Metformin Group (MG)
Drug: Placebo — Placebo oral tablets. Prescribed: Once daily PO with meals and 200 mL of water.
  Arms: The Placebo Control Group (PCG)

SUMMARY:
The aim of this multicenter, pragmatic, open-label, randomized, placebo-controlled clinical trial is to test whether repurposing metformin for the treatment of atrial fibrillation will be effective in decreasing patients' hospitalization, adverse major cardiovascular events, and non-cancer death.

Participants will be randomized into 2 study arms (385 participant each), whereby:

* The Metformin Group (MG): will receive metformin oral tablets in addition to the standard rate/rhythm control strategy and anticoagulation.
* The Placebo Control Group (PCG): will receive placebo oral tablets as a control group in addition to the standard rate/rhythm control strategy and anticoagulation.

Then both arms will be compared according to the these endpoints:

* The primary endpoint is hospitalization due to an episodic AF or an AF with a rapid or slow ventricular response (in the case of permanent AF).
* The secondary endpoint is a composite of non-fatal major cardiovascular adverse events or non-cancer death.

The non-fatal major cardiovascular adverse events include:

* Hospitalization due to heart failure.
* Non-fatal myocardial infarction.
* Non-fatal stroke.
* Hospitalization due to unstable angina.

DETAILED DESCRIPTION:
* Type of The Study: Interventional, Placebo-Controlled Clinical Trial.
* Therapeutic Area: Cardiology, Arrhythmia.
* Purpose: Treatment.
* Aim: Whether repurposing metformin for the treatment of atrial fibrillation will be effective in decreasing patients' hospitalization, adverse major cardiovascular events, and non-cancer death.
* Assignment: Parallel.
* Allocation: Randomized.
* Masking: Pragmatic, Open-Label.
* Duration: 12 months of follow-up.
* Rationale: Atrial fibrillation (AF) is the most common heart arrhythmia [1], in which atria contract rapidly and irregularly and the contraction of atria and ventricles is no longer coordinated. Current guidelines for the treatment of AF recommend medication to avoid blood clotting and stroke, control heart rate, and restore sinus rhythm. However, the available treatments show limited efficiency and may have side effects associated with increased morbidity and mortality [2], emphasizing an urgent need for new or repurposed therapies. Lal and colleagues [3] reported an integrative approach-combining transcriptomics, iPSCs, and epidemiological evidence-to identify and repurpose metformin, a main first-line medication for the treatment of type 2 diabetes, as an effective risk reducer for atrial fibrillation. Interestingly, metformin enhances the life span in invertebrate and vertebrate laboratory models [4], and similar gene-expression-based drug-repurposing studies targeting aging identified metformin, among others, as a pro-longevity agent [5]. Diabetes and AF are both age-associated and often co-morbid conditions. Metformin is being tested in the Targeting Aging with Metformin (TAME) trial [6] to develop effective next-generation drugs to increase healthspan and lifespan. Additionally, metformin seems to be associated with a lower risk of atrial fibrillation and ventricular arrhythmias as compared with another anti-diabetic drug category which is sulfonylureas [7]. The potential antiarrhythmic role of metformin in patients with AF could be due to the effects of metformin on preventing the structural and electrical remodeling of the left atrium via attenuating intracellular reactive oxygen species, activating 5' adenosine monophosphate-activated protein kinase, improving calcium homeostasis, attenuating inflammation, increasing connexin-43 gap junction expression, and restoring small conductance calcium-activated potassium channels current [8]. Despite the solid preclinical, integrative, and retrospective analyses, the effect of metformin on patients with AF regarding morbidity and mortality has not be established using a perspective, randomized, controlled trial.
* Inclusion Criteria: Age more than 20 years and less than 65 years, willing and able to provide written informed consent prior to performing study procedures, and diagnosed by atrial fibrillation (first detected, paroxysmal, persistent, longstanding persistent, or permanent).
* Exclusion Criteria: Critically-ill patients who are admitted to ICU, advanced congestive heart failure, liver cell failure, chronic kidney disease with eGFR <45 mL/min/1.73 m², diabetic ketoacidosis with or without coma, concomitant treatment with carbonic anhydrase inhibitors, septicemia, shock, hypoxia, dehydration, blood dyscrasias, pregnancy, lactation, chronic muscle diseases, acute trauma or burns within 2 weeks, and history of allergy to the implemented drugs.
* Methods: 770 enrolled AF patients who are candidates for metformin treatment according to the study criteria at the time of presentation, will undergo the following at the time of enrollment and during the bimonthly follow-ups:

  * General and Local cardiac examination.
  * CBC.
  * Chemistry Panel including KFTs, LFTs.
  * Serum electrolytes levels.
  * Resting surface 12 leads ECG.
  * Baseline echocardiography.
* Interventions:

  * Drug: metformin 850 mg oral tablets. Prescribed: Once daily PO with meals and 200 mL of water. The dose can be up-titrated to 1500-2000 mg divided q8-12hr with meals in enrolled diabetic patients as a monotherapy or combined with sulfonylurea.

Other Name: Glucophage.

* Drug: Placebo oral tablets. Prescribed: Once daily PO with meals and 200 mL of water. Other Name: Placebo

  - Study Arms:
* The Metformin Group (MG): 385 patients will receive metformin oral tablets in addition to the standard rate/rhythm control strategy and anticoagulation.
* The Placebo Control Group (PCG): 385 patients will receive placebo oral tablets as a control group in addition to the standard rate/rhythm control strategy and anticoagulation.

Endpoints:

* The primary endpoint is hospitalization due to an episodic AF or an AF with a rapid or slow ventricular response (in the case of permanent AF).
* The secondary endpoint is a composite of non-fatal major cardiovascular adverse events or non-cancer death.

The non-fatal major cardiovascular adverse events include:

* Hospitalization due to heart failure.
* Non-fatal myocardial infarction.
* Non-fatal stroke.
* Hospitalization due to unstable angina.

  • Safety: In terms of safety, a composite of metformin side effects comprising GIT symptoms, hypoglycemia, and lactic acidosis will be considered.
* Ethics: The study will be conducted in compliance with human studies committees' regulations of the authors' institutions and COPE guidelines, including patient consent as appropriate.
* Competing Interests: The authors will declare any commercial or financial relationships that could be construed as a potential conflict of interest.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written informed consent prior to performing study procedures.
* Atrial fibrillation (first detected, paroxysmal, persistent, longstanding persistent, or permanent)*.

  * Types of atrial fibrillation:
* First detected: only one diagnosed episode.
* Paroxysmal: recurrent episodes that stop on their own in less than seven days.
* Persistent: recurrent episodes that last more than seven days.
* Longstanding persistent: recurrent episodes that last more than twelve months.
* Permanent: atrial fibrillation that has been accepted, and for which a solely rate control strategy has been decided upon.

Exclusion Criteria:

* Critically-ill patients who are admitted to ICU.
* Advanced congestive heart failure.
* Liver cell failure.
* Chronic kidney disease with eGFR <45 mL/min/1.73 m².
* Diabetic ketoacidosis with or without coma.
* Concomitant treatment with carbonic anhydrase inhibitors.
* Septicemia.
* Shock.
* Hypoxia.
* Dehydration.
* Blood Dyscrasias.
* Alcoholism.
* Pregnancy.
* Lactation.
* Chronic muscle diseases.
* Acute trauma or burns within 2 weeks.
* History of allergy to the implemented drugs.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 770 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2025-01 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Primary Endpoint | 12 months since randomization
  The primary endpoint is hospitalization due to an episodic AF or an AF with a rapid or slow ventricular response (in the case of permanent AF).

SECONDARY OUTCOMES:
Secondary Endpoint | 12 months since randomization
  The secondary endpoint is a composite of non-fatal major cardiovascular adverse events or non-cancer death.
  The non-fatal major cardiovascular adverse events include:
  * Hospitalization due to heart failure.
  * Non-fatal myocardial infarction.
  * Non-fatal stroke.
  * Hospitalization due to unstable angina.

CONTACTS AND LOCATIONS:
Overall Officials: Eslam Abbas, MBBCh, MSC, Principal Investigator — Arab Contractors Medical Centre, and Dar El Salam Cancer Center
Locations (1):
- Arab Contractors Medical Centre, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Data can be shared with researchers who submit a proposal with a valuable research question as assessed by the clinical research office of Al-Azhar University. Requests should be directed to the corresponding authors.
Supporting Information: Study Protocol, SAP
Time Frame: Data that underlie the results reported in this study will be available upon publication.
Access Criteria: Data can be shared with researchers who submit a proposal with a valuable research question.

REFERENCES:
- [Background] Chung MK, Eckhardt LL, Chen LY, Ahmed HM, Gopinathannair R, Joglar JA, Noseworthy PA, Pack QR, Sanders P, Trulock KM; American Heart Association Electrocardiography and Arrhythmias Committee and Exercise, Cardiac Rehabilitation, and Secondary Prevention Committee of the Council on Clinical Cardiology; Council on Arteriosclerosis, Thrombosis and Vascular Biology; Council on Cardiovascular and Stroke Nursing; and Council on Lifestyle and Cardiometabolic Health. Lifestyle and Risk Factor Modification for Reduction of Atrial Fibrillation: A Scientific Statement From the American Heart Association. Circulation. 2020 Apr 21;141(16):e750-e772. doi: 10.1161/CIR.0000000000000748. Epub 2020 Mar 9. PMID 32148086
- [Background] Schwaerzer G. Repurposing metformin for treatment of atrial fibrillation. Nat Cardiovasc Res. 2022 Nov;1(11):972. doi: 10.1038/s44161-022-00170-1. No abstract available. PMID 39195908
- [Background] Lal JC, Mao C, Zhou Y, Gore-Panter SR, Rennison JH, Lovano BS, Castel L, Shin J, Gillinov AM, Smith JD, Barnard J, Van Wagoner DR, Luo Y, Cheng F, Chung MK. Transcriptomics-based network medicine approach identifies metformin as a repurposable drug for atrial fibrillation. Cell Rep Med. 2022 Oct 18;3(10):100749. doi: 10.1016/j.xcrm.2022.100749. Epub 2022 Oct 11. PMID 36223777
- [Background] Vinciguerra M, Olier I, Ortega-Martorell S, Lip GYH. New use for an old drug: Metformin and atrial fibrillation. Cell Rep Med. 2022 Dec 20;3(12):100875. doi: 10.1016/j.xcrm.2022.100875. PMID 36543101
- [Background] Donertas HM, Fuentealba Valenzuela M, Partridge L, Thornton JM. Gene expression-based drug repurposing to target aging. Aging Cell. 2018 Oct;17(5):e12819. doi: 10.1111/acel.12819. Epub 2018 Aug 9. PMID 29959820
- [Background] Barzilai N, Crandall JP, Kritchevsky SB, Espeland MA. Metformin as a Tool to Target Aging. Cell Metab. 2016 Jun 14;23(6):1060-1065. doi: 10.1016/j.cmet.2016.05.011. PMID 27304507
- [Background] Ostropolets A, Elias PA, Reyes MV, Wan EY, Pajvani UB, Hripcsak G, Morrow JP. Metformin Is Associated With a Lower Risk of Atrial Fibrillation and Ventricular Arrhythmias Compared With Sulfonylureas: An Observational Study. Circ Arrhythm Electrophysiol. 2021 Mar;14(3):e009115. doi: 10.1161/CIRCEP.120.009115. Epub 2021 Feb 7. PMID 33554609
- [Background] Nantsupawat T, Wongcharoen W, Chattipakorn SC, Chattipakorn N. Effects of metformin on atrial and ventricular arrhythmias: evidence from cell to patient. Cardiovasc Diabetol. 2020 Nov 24;19(1):198. doi: 10.1186/s12933-020-01176-4. PMID 33234131